CLINICAL TRIAL: NCT06978517
Title: Effect of Postural Stability System Comparison to Nintendo Wii Fit Balance Training on Fall Risk and Postural Stability in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/73
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Fall Risk; Postural Stability; Balance; Elderly
Keywords: Fall risk; postural stability; Biodex balance system; Nintendo Wii fit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodex balance system (Experimental): It includes the following techniques for training: weight shift training, limits of stability, and weight training techniques It includes 15 participants and includes warm-up and cool-down period
  Interventions: Procedure: Biodex balance system
- Nintendo Wii fit (Active Comparator): Nintendo Wii Fit Balance Training, which includesthe following games:
  * table tilt
  * ski slalom
  * Penguin slide
  * Tightrope walk
  * Soccer heading
  * Balance bubble It includes 15 participants and playing each game for 10 minutes
  Interventions: Procedure: nintendo Wii fit balance training

INTERVENTIONS:
Procedure: Biodex balance system — Participants assigned to the Biodex balance training group underwent balance rehabilitation using the Biodex Balance System SD, a computerized platform designed to assess and train postural stability. Each participant engaged in training sessions three times per week, with each session lasting approximately 30 minutes, over a total period of six weeks. The intervention began with exercises conducted on a higher stability level (e.g., Level 8), gradually progressing to lower stability levels (e.g., Level 2) to increase the challenge as participants' balance improved. The training included both static and dynamic tasks aimed at enhancing weight shifting, center-of-gravity control, and response to instability. Real-time visual biofeedback was provided via the system's screen, enabling participants to monitor their performance and maintain motivation. All sessions were conducted under the supervision of a qualified physiotherapist to ensure proper technique and safety.
  Arms: Biodex balance system
Procedure: nintendo Wii fit balance training — Participants in the Nintendo Wii Fit training group engaged in balance exercises using the Nintendo Wii console and Wii Fit balance board. This interactive system includes a variety of balance-focused activities and games that simulate real-life balance challenges in a virtual environment. The training was conducted three times per week, with each session lasting approximately 30 minutes, over a six-week period. Exercises included selected Wii Fit balance games (such as Ski Slalom, Table Tilt, and Tightrope Walk) and yoga-based poses (such as Tree Pose and Warrior), which encouraged participants to engage their core and lower limb muscles while maintaining postural alignment. The difficulty level was gradually increased by introducing more complex tasks and longer balance durations as participants progressed. The system provided immediate visual and auditory feedback, allowing users to track their scores and improvements in real time. All sessions were performed under supervision.
  Arms: Nintendo Wii fit

SUMMARY:
Human balance is a complex multidimensional concept related to postural control, and it refers essentially to the ability to maintain a posture (e.g., sitting or standing), move between postures, and not fall when reacting to an external disturbance. One-third to one-half of the population over age 65 reports some difficulty with balance or ambulation .Because of the high incidence of balance and mobility disorders in older adults, interventions are necessary that optimize the performance of balance- and mobility-related activities older adults .

The aim of the current study will benefit clinicians and physiotherapists as it provide an insight to the benefits of balance training. The practical application of balance training will provide neurological advantages tothe geriatric population to allow lesser fall risk and postural instability.

The study will be a non-blinded randomized control trial, consisting of two groups. Study will be conducted over 1 year. Subjects will be selected via a non-probability purposive sampling technique using a coin toss method, followed by randomization into two groups (A and B). Ethical approval will be obtained from the ERC FUMC. One group will receive Nintendo Wii Fit balance training while the second group will receive postural stability system training over 8 weeks. Baseline tests will be performed before and after the intervention for balance, postural stability, and sensory integration. Data will be entered and analyzed on SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* Age 55years and above
* Males and females both
* Berg balance scale score 21-40
* TUG in less than 20 sec

Exclusion Criteria:

* Use of a wheelchair or walker.
* Any diagnosed neurological condition.
* Any severe musculoskeletal condition.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Balance | 8 weeks
  Berg balance scale is used to assess functional balance and mobility, particularly in the elderly and those with balance impairment. It's a 14-item scale where each item is scored on a 5-point scale (0-4), with a total score ranging from 0 to 56. The higher the score, the better the patient's balance
Fall risk | 8 weeks
  The Timed Up and Go (TUG) test is a simple and widely used assessment of fall risk that measures the time it takes for someone to rise from a chair, walk a certain distance (usually 3 meters), turn around, and walk back to sit down.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan